CLINICAL TRIAL: NCT01765140
Title: Treatment Use of 3,4-Diaminopyridine in Congenital Myasthenic Syndrome
Brief Title: Treatment Use of 3,4-Diaminopyridine
Status: No longer available | Type: Expanded Access
Sponsor: Vern C. Juel, M.D. (Other)
Responsible Party: Sponsor-Investigator, Vern C. Juel, M.D., Professor of Neurology, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00007811
Record Dates: First submitted 2013-01-06; First posted 2013-01-10 (Estimated); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Myasthenic Syndromes, Congenital
Keywords: 3,4 diaminopyridine (DAP)
MeSH Terms: conditions — Myasthenic Syndromes, Congenital | interventions — Amifampridine

INTERVENTIONS:
Drug: 3,4-diaminopyridine — Treatment use of 3,4-DAP for patients with congenital myasthenic syndrome (CMS)
  Other Names: DAP

SUMMARY:
This protocol provided 3,4 diaminopyridine (DAP) under a treatment-use IND to patients with congenital myasthenic syndrome (CMS). It is now closed.

DETAILED DESCRIPTION:
CMS diagnoses were made based on clinical, electrophysiologic and molecular genetic findings. All patients were referred to the PI for DAP treatment. This study enrolled minors and adults.

CMS patients under age 18 years were included if their parent or guardian gave written permission. Minors who turned 18 while in the program were re-consented as adults.

The dose of DAP was determined individually for each patient. Adults were started with a dose of 10 mg 3-4 times daily, increased over several weeks to the dose that produced the maximum symptomatic response, not to exceed 100 mg daily. Pyridostigmine bromide (PB) was often added at low doses and increased to the dose that produced the best response, not to exceed 360 mg daily. In children, equivalent doses of these medications were calculated on a surface area basis. The doses of DAP and PB were periodically adjusted to assure that the smallest effective doses are used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of congenital myasthenic syndrome (CMS)
* Women of childbearing potential must have negative pregnancy test and agree to practice adequate contraception while taking DAP
* Must be competent to give consent

Exclusion Criteria:

* Known seizure disorder
* Pregnancy
* Known cardiac arrhythmia or evidence of significant arrhythmia on screening ECG
* Known hepatic, renal or hematologic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Vern C. Juel, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Background] Sanders DB, Juel VC, Harati Y, Smith AG, Peltier AC, Marburger T, Lou JS, Pascuzzi RM, Richman DP, Xie T, Demmel V, Jacobus LR, Ales KL, Jacobus DP; Dapper Study Team. 3,4-diaminopyridine base effectively treats the weakness of Lambert-Eaton myasthenia. Muscle Nerve. 2018 Apr;57(4):561-568. doi: 10.1002/mus.26052. Epub 2018 Feb 2. PMID 29280483